CLINICAL TRIAL: NCT01375569
Title: A Phase II Study of TRC105 in Patients With Hepatocellular Carcinoma (HCC) Who Have Progressed on Sorafenib
Brief Title: TRC105 for Liver Cancer That Has Not Responded to Sorafenib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110181; 11-C-0181
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Carcinoma, Hepatocellular
Keywords: CD105; Monoclonal Antibody; Anti-Angiogenic; Chimeric; Apoptosis; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TRC105 in Liver Cancer (Experimental): TRC105 is an experimental cancer drug designed to slow or stop the growth of tumors. It does this by preventing the growth of new blood vessels that feed these tumors. This drug is being used to test the safety and effectiveness to treat liver cancer that has not responded to standard therapy. TRC105 will be given as an intravenous infusion every two weeks.
  Interventions: Drug: TRC105

INTERVENTIONS:
Drug: TRC105

SUMMARY:
Background:

- TRC105 is an experimental cancer drug. It is designed to slow or stop the growth of tumors. It does this by preventing the growth of new blood vessels that feed these tumors. People with hepatocellular carcinoma (or liver cancer) sometimes do not respond to standard treatments. This includes the cancer drug sorafenib.

Objectives:

- To test the safety and effectiveness of TRC105 to treat liver cancer that has not responded to standard therapy.

Eligibility:

* People at least 18 years of age who have hepatocellular carcinoma (or liver cancer) that has not responded to standard therapy. Participants also will not be eligible for a liver transplant.
* No anticoagulation therapy is allowed with the exception of low-dose aspirin.
* No history of bleeding disorders, peptic ulcer disease or gastritis.

Design:

* Participants will have a physical exam and medical history. They will also have blood and urine tests, and imaging studies.
* Participants will receive TRC105 once a week. They will also have two daily doses of a steroid the day before each treatment. This will help prevent known side effects.
* Participants will be monitored with blood and urine tests. They will also have imaging studies every two months to study the effect of the drug on tumor growth.
* Participants will continue to have TRC105 as long as they do not have severe side effects and their liver cancer stops growing or shrinks. After stopping TRC105, they will have yearly visits with physical exams and blood tests.

DETAILED DESCRIPTION:
Background:

* Worldwide, hepatocellular carcinoma (HCC) is the fifth most common malignancy with a median survival of 6-9 months. The Study of Heart and Renal Protection (SHARP) study established Sorafenib as a standard consideration in this disease and set the bar for future studies of systemic therapy. There is no standard therapy for patients whose disease has progressed despite Sorafenib therapy.
* TRC105 is a chimeric, anti-angiogenic monoclonal antibody that binds CD105, a transmembrane receptor overexpressed by proliferating endothelial cells. TRC105 binds to CD105-expressing endothelial cells and mediates growth inhibition, apoptosis and antibody-dependent cell-mediated cytotoxicity (ADCC).

Objectives:

Primary:

-To evaluate time to tumor progression (TTP) for TRC105 in HCC.

Secondary:

* To evaluate safety of TRC105 in HCC.
* To evaluate the immunogenicity of TRC105 as measured by human antichimeric antibody (HACA) and human antimouse antibody formation.
* To evaluate anti-tumor response as determined by standard and European Association for the Study of the Liver (EASL) -modified Response Evaluation Criteria in Solid Tumors (RECIST) response criteria.
* To perform correlative studies assessing potential biomarkers of response to TRC105.

Eligibility:

* Histologically or cytologically confirmed diagnosis of HCC.
* Childs-Pugh A or B (7 points) cirrhosis only is allowed.
* Patients must have disease that is not amenable to potentially curative resection.
* Patients must have progressed on or been intolerant of prior sorafenib therapy.
* No history of bleeding varices (unless subsequent liver transplant). All patients must have had endoscopic evaluation within 6 months of starting study.
* No history of bleeding varices in previous 1 year (unless subsequent liver transplant). No anti-coagulation (except low-dose aspirin).

Design:

* This is a single-arm phase II study of TRC105 in patients with HCC.
* TRC105 will be administered as an intravenous infusion every two weeks. Patients will be re-staged every 8 weeks.
* The primary endpoint of the study will be Time to Tumor Progression (TTP). The primary purpose of this study is to evaluate the ability of TRC105 as a second line treatment to improve upon the time to progression (TTP) of patients with refractory HCC.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of Hepatocellular Carcinoma (HCC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study.

Or

histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC.

* Patients must have disease that is not amenable to potentially curative resection or ablative techniques. In addition, disease must not be amenable to transhepatic arterial chemoembolization (TACE). Patients may have had prior TACE and had disease progression following it. Patients must not be considered potential candidates for liver transplantation. This determination will be made after hepatobiliary surgical input at the NCI multidisciplinary conference.
* All patients enrolled will be required to have measurable disease.
* If liver cirrhosis is present, patient must have a Child-Pugh A classification.
* Patients must have progressed on or been intolerant of prior sorafenib therapy.
* Patients must with cirrhosis have had esophagogastric endoscopy within the previous 6 months prior to study entry for the assessment of varices. If the patient has not had this done they must be willing to undergo this procedure prior to study entry.
* Age greater than or equal to 18 years
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/mcL
  * Platelets greater than or equal to 60,000/mcL
  * Total bilirubin less than or equal to 3 times upper normal limits
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 10 times upper limit of normal
  * Creatinine less than or equal to 1.5 times upper normal limits OR creatinine clearance greater than or equal to 40 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal, as calculated by the Cockcroft Gault formula.
* Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
* Patients must not have other invasive malignancies within the past 3 years (with the exception of non-melanoma skin cancers, carcinoma in situ of the cervix and noninvasive bladder cancer).
* Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment.
* Patient must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy, large field radiotherapy, or major surgery must wait 4 weeks prior to entering the study (2 weeks is sufficient for targeted systemic therapy provided toxicity has recovered to less than or equal to grade 1).
* Patients may not be receiving any anti-cancer agents not approved by the Food and Drug Administration (FDA) within the past 4 weeks.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Proteinuria, as demonstrated by a 24 hour protein of greater than or equal to 2000 mg. Urine protein will be screened by urine protein-creatinine ratio (UPC). For urine protein-to-creatinine (UPC) ratio > 1.0, a 24-hour urine protein will need to be obtained and the level should be < 2000 mg for patient enrollment.
* Uncontrolled intercurrent illness including, but not limited to, hypertension (systolic blood pressure (BP) 160, diastolic BP > 100), ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* No anti-coagulation therapy is allowed with the exception of low-dose aspirin.
* No bleeding diathesis.
* Patients with a history of bleeding varices in previous 1 year are excluded (unless patient has subsequently had a liver transplant). Those with gastric varices or varices that are deemed as high risk by the endoscopist should be placed on appropriate medical therapy as advised by the gastroenterologist.
* History of peptic ulcer disease or hemorrhagic gastritis within 6 months of TRC105 administration, unless patient has received adequate treatment for peptic ulcer disease or hemorrhagic gastritis and has evidence of complete resolution documented by esophagogastroduodenoscopy (EGD). Mild gastritis is allowed.
* Corrected QT interval (QTc) > 500 msec.
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and TRC105. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that TRC105 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to TRC105.
* History of hypersensitivity reaction to human or mouse antibody products.
* Patients with a history of familial bleeding disorders.
* Patients with a history of hereditary hemorrhagic telangiectasia (Osler-Weber-Rendu syndrome).
* Pregnancy and breast feeding are exclusion factors. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment.

INCLUSION OF WOMEN AND MINORITIES:

-Men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-06-22 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2015-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Yoo HY, Patt CH, Geschwind JF, Thuluvath PJ. The outcome of liver transplantation in patients with hepatocellular carcinoma in the United States between 1988 and 2001: 5-year survival has improved significantly with time. J Clin Oncol. 2003 Dec 1;21(23):4329-35. doi: 10.1200/JCO.2003.11.137. Epub 2003 Oct 27. PMID 14581446
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0181.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRC105 in Liver Cancer
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TRC105 in Liver Cancer
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.46 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression (TTP) for TRC105 in Hepatocellular Carcinoma (HCC).
Description: Time to tumor progression is defined as the proportion of participants who are progression free after 4 months on study. Progression is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 2 years
Measure: Mean (Full Range); unit: Weeks
Arm/Group | TRC105 in Liver Cancer
Number analyzed (Participants) | 11
Weeks | 12 [4 to 32]

2. Secondary Outcome: Count of Participants With Adverse Events
Description: here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 25 months, 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 in Liver Cancer
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: 25 months, 15 days
Arm/Group | TRC105 in Liver Cancer
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 in Liver Cancer (N=11)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) — This adverse event is not related to the TRC105 study drug.
Hepatic failure (Hepatobiliary disorders) | 1 (1) — This adverse event is not related to the TRC105 study drug.
Lung infection (Infections and infestations) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — malignant neoplasm
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 in Liver Cancer (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 4 (6)
Alanine aminotransferase increased (Investigations) | 6 (13)
Alkaline phosphatase increased (Investigations) | 8 (14)
Anemia (Blood and lymphatic system disorders) | 7 (23)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 9 (27)
Blood bilirubin increased (Investigations) | 9 (19)
Blurred vision (Eye disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Investigations) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema limbs (General disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Eye disorders - Other, specify (eye itchiness and redness) (Eye disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 2 (5)
Flushing (Vascular disorders) | 1 (1)
Gallbladder infection (Infections and infestations) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (15)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (20)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 7 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Infections and infestations - Other, specify (oral thrush) (Infections and infestations) | 2 (2)
Infusion related reaction (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (3)
Oral hemorrhage (Gastrointestinal disorders) | 3 (5)
Pain (General disorders) | 4 (9)
Platelet count decreased (Investigations) | 5 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (hemoptysis) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Serum amylase increased (Investigations) | 2 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No